CLINICAL TRIAL: NCT00468520
Title: A Prospective, Randomized Trial of Transcervical Foley Catheter With or Without Oxytocin for Preinduction Cervical Ripening
Brief Title: Adjuvant Oxytocin for Preinduction Ripening With a Foley catheter--a Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 20030859
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Pregnancy; Induced Labor; Cervical Ripening
Keywords: induction of labor; cervical ripening; Foley catheter; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: low dose oxytocin

SUMMARY:
The transcervical Foley catheter (TFC) is a proven and effective mode of cervical ripening. It is common practice to use TFC with simultaneous low-dose oxytocin under the assumption that the combination results in a more successful labor induction. Scientific validation of this practice is lacking. We seek to determine if the addition of oxytocin to TFC improves induction success.

DETAILED DESCRIPTION:
This is a prospective, randomized trial that aims to enroll 200 singleton pregnancies presenting for preinduction ripening. Patients will be randomized to receive either TFC alone (control) or TFC plus low-dose oxytocin (treatment). Providers will not blinded to use of oxytocin and labor was managed according to routine obstetric protocols. This study is powered to detect a 20% difference in the proportion of patients delivered within 24 hours, the primary outcome. Secondary outcomes are related to vaginal delivery rate, duration of induction, complications, and pain management.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* presenting for induction as determined by their primary obstetrical provider
* with fetuses in cephalic presentation
* gestational age greater than 23 weeks

Exclusion Criteria:

* any condition precluding vaginal delivery
* estimated fetal weight >4500 grams
* a previous attempt at ripening or induction during the pregnancy
* clinically significant cervical or vaginal infection
* chorioamnionitis
* HIV
* hepatitis B or C
* unexplained vaginal bleeding
* low-lying placenta
* abnormal cervical anatomy or cervical cerclage
* latex allergy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2003-11; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Delivery rate (proportion) | Within 24 hours

SECONDARY OUTCOMES:
vaginal delivery rate | within 24 hours
use of anesthesia/analgesia | during induction and labor
overall complication rate (composite)
duration of induction and labor

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Devine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515